CLINICAL TRIAL: NCT00060138
Title: A Phase I-II, 24-Week, Multi-Center, Double-Blind, Randomized, Dose-Ranging Study To Evaluate The Safety And Efficacy Of A Humanized Monoclonal Antibody To PTHrP Versus Zoledronic Acid In Patients With Breast Cancer Metastatic To Bone
Brief Title: Monoclonal Antibody Compared With Zoledronate in Treating Women With Breast Cancer and Bone Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CWRU-080235; CDR0000299530 (Registry Identifier: PDQ (Physician Data Query)); CBI-1102; CBI-CAL-03
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Hypercalcemia of Malignancy; Metastatic Cancer; Pain
Keywords: hypercalcemia of malignancy; stage IV breast cancer; recurrent breast cancer; bone metastases; pain
MeSH Terms: conditions — Breast Neoplasms; Humoral Hypercalcemia Of Malignancy; Neoplasm Metastasis; Pain | interventions — Antibodies, Monoclonal; Zoledronic Acid

INTERVENTIONS:
Biological: monoclonal antibody CAL
Drug: zoledronic acid

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Zoledronate may prevent bone loss and stop the growth of tumor cells in bone. It is not yet known whether monoclonal antibody is more effective than zoledronate in treating women who have breast cancer and bone metastases.

PURPOSE: Randomized phase I/II trial to compare the effectiveness of monoclonal antibody with that of zoledronate in treating women who have breast cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and tolerability of monoclonal antibody CAL vs zoledronate in women with breast cancer and bone metastases.
* Compare, preliminarily, the potential effects of these drugs on skeletal events/manifestations related to bone metastases, including hypercalcemia, bone pain, bone metastatic lesions, complications (e.g., pathologic fracture and spinal cord compression), and interventions (e.g., surgery and radiotherapy) in these patients.
* Compare changes in ECOG performance status in patients treated with these drugs.
* Determine the pharmacokinetics of monoclonal antibody CAL in these patients.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to average prestudy pain score on question 3 of a daily electronic telephone pain diary (less than 3 vs 3 or more) and prior bisphosphonate therapy (yes vs no). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive monoclonal antibody CAL IV over 30-60 minutes on day 1.
* Arm II: Patients receive a lower dose of monoclonal antibody CAL as in arm I.
* Arm III: Patients receive a lower dose (lower than arm II) of monoclonal antibody CAL as in arm I.
* Arm IV: Patients receive zoledronate IV over 30-60 minutes on day 1. Treatment in all arms repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients keep a pain diary throughout study participation.

Patients are followed at 24 weeks.

PROJECTED ACCRUAL: A total of 72 patients (18 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer
* Radiographical evidence of at least 1 bone metastasis

  * No prior radiotherapy or surgery to bone metastasis
  * No radiotherapy or surgery anticipated for bone metastasis within the next 24 weeks
* Bone pain severity score of at least 1 on 5 of 7 days as determined by question 3 of the Brief Pain Inventory (BPI)
* No bone metastases to a weight-bearing bone at imminent risk for pathologic fracture or surgical intervention
* No vertebral metastases that place the patient at imminent risk of spinal cord compression
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Pre- or post-menopausal

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* WBC at least 2,000/mm^3
* Lymphocyte count at least 500/mm^3
* Granulocyte count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic

* ALT or AST no greater than 2.5 times upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN

Renal

* Calcium no greater than 10.1 mg/dL
* No oliguria, defined as less than 30 mL urine per 2-hour collection
* No acute renal failure
* Creatinine no greater than 2.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No sepsis
* No known or anticipated contraindication to study drugs

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 weeks since initiation of a new chemotherapy regimen

Endocrine therapy

* More than 3 weeks since initiation of a new hormonal therapy regimen

Radiotherapy

* See Disease Characteristics
* More than 3 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* More than 60 days since prior bisphosphonates
* More than 30 days since prior investigational drugs
* No change in analgesic drug regimen during the screening period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Silverman, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States